CLINICAL TRIAL: NCT00428987
Title: Study of the Phenotype of Overweight and Obese Adults
Brief Title: Physical and Behavioral Traits of Overweight and Obese Adults
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070077; 07-DK-0077
Record Dates: First submitted 2007-01-27; First posted 2007-01-30 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01-05

CONDITIONS: Obesity; Healthy Volunteers
Keywords: Energy Expenditure; Body Composition; Obesity; Metabolism; Phenotype; Natural History; Morbid Obesity; Overweight; Healthy Volunteer
MeSH Terms: conditions — Obesity; Obesity, Morbid; Overweight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- lean: Normal weight men and women over the age of 18 years with BMI greater than 18.5 and less than 25, who are reasonably healthy
- obese: Obese men and women over the age of 18 years with BMI greater than 30, who are reasonably healthy
- overweight: Overweight men and women over the age of 18 years with BMI greater than 25 and less than 30, who are reasonably healthy

SUMMARY:
This study will describe the phenotype (physical and behavioral traits) of overweight and obese people. It will characterize the hormones, metabolism, food preferences, fitness and physical activity levels, sleep patterns and thought processes in people with and without weight problems. Genetic material will be collected for studies of the internal codes that influence body weight.

People over 18 years of age from all weight categories (lean, overweight, obese) who are reasonably healthy may be eligible for this study. Participants undergo the following tests and procedures:

* Physical exam, electrocardiogram, blood and urine tests, instructions for recording food intake for 7 days
* Metabolic studies for menstruating women.
* Resting metabolic rate to study how many calories the body burns at rest.
* Mixed meal test to measure hormones such as insulin that regulate blood sugar.
* Glucose tolerance test to determine how sensitive the body is to insulin.
* 24-hour energy expenditure to measure the amount of oxygen breathed in and the amount of carbon dioxide breathed out.
* Repeat 24-hour energy expenditure.
* Diurnal blood sampling and temperature assessment to study the body s internal clock.
* Air-displacement plethysmography (Bod Pod) to measure body composition.
* Dual energy x-ray absortiometry (DEXA) to measure body fat and bone density.
* Repeat Bod Pod and DEXA.
* Anthropometric measurements and bioelectrical impedance to measure height, weight, and circumferences, skinfold thickness, fluid status and percentage body fat.
* Bromide dilution to measure the amount of water not in cells in the body.
* Doubly labeled water to measure the amount of calories burned in a 7-day period.
* 24-hour diet reports.
* Endothelial reactivity to measure how the blood vessels stretch or dilate for assessing cardiovascular health.
* Treadmill or bicycle exercise capacity test.
* Physical activity monitor.
* Unicorder to detect any breathing difficulties that may interfere with sleep.
* Fat and muscle biopsy to look for variations in gene expression in fat tissue and muscle.
* Neurocognitive testing to check memory, decision-making, hand-eye coordination, and reasoning.
* Evaluation of mood problems and assess personality type.
* Evaluation to assess the quantity and quality of pain experienced.
* Taste testing to determine the response to bitter, salty, sweet and sour substances.
* Occupational therapy evaluation to explore the subject's adaptations, if any, for performing personal, social or professional activities; the subject's views on his or her weight, body size and shape, and strategies to control weight.

DETAILED DESCRIPTION:
Although complex metabolic, hormonal, and neural networks operate to control body weight, obesity is in most cases, the result of over-feeding and inactivity. In most obese patients, patterns of fundamental behavior determine the success or failure of weight loss interventions. Behavior is controlled to some degree by conscious decision making and is influenced by signals from the integrated networks involved in body weight regulation. The contributions of behavior, environment, socioeconomic status, physiology and genetics assure that no single therapeutic regimen will be successful in all obese individuals. In order to explore the factors that impede weight loss and result in weight regain, the obese phenotype and its variants must be defined. The purpose of this study is to detail hormonal, metabolic, cognitive and behavioral traits across the spectrum of weight categories utilizing the state-of the-art facilities of the Metabolic Units at the Mark O. Hatfield Clinical Research Center, NIH. Genetic material will be banked for analysis of phenotypic subgroups as they emerge.

Patients over the age of 18 are eligible for this study. While childhood obesity is an important public health issue, the variables of growth and hormonal controls will be delineated in separate studies. Over-weight and obese patients are encouraged to participate in as full an evaluation as feasible. Lean individuals will be recruited to create a normative database for body composition (dual energy x-ray absortiometry, air displacement plethysmography), energy expenditure (resting energy expenditure, 24h respiratory chamber and doubly labeled water) and other techniques used to study traits of importance. The study will be conducted in both the inpatient and outpatient setting and can include evaluation of hormones, diurnal variation, sleep, eating behavior and taste perception, physical fitness, psychological and neurocognitive functioning. Importantly, this protocol is the means by which pilot data are obtained to develop novel approaches and hypotheses for studying obesity and its associated traits.

ELIGIBILITY:
* INCLUSION CRITERIA:

Obese subjects:

1. Obese men and women over the age of 18 years
2. BMI > 30

Overweight subjects:

1. Overweight men and women over the age of 18 years
2. BMI > 25 and < 30

Control subjects (may be matched for age, sex and years of education):

1. Normal weight men and women over the age of 18 years
2. BMI > 18.5 and < 25

EXCLUSION CRITERIA:

1. Patients with significant physical limitations that may preclude them from completing the majority of the tests in this study
2. Current unstable medical conditions including cardiac ischemia, severe respiratory insufficiency requiring oxygen therapy, hepatic or cardiac failure as assessed by history and physical exam
3. Any psychiatric condition that would preclude participation in the study
4. Patients unwilling or unable to give informed consent
5. Pregnant woman.

Additional exclusion for lean control subjects:

1. Previous history of obesity as an adolescent or adult
2. Current or past history of eating disorders such as anorexia nervosa or bulimia

The NIH Patient Recruitment and Public Liaison Office will receive inquiries from interested study subjects. Pre-screening by this office will exclude patients who require more than minimal assistance to complete activities of daily living in order to select subjects who can safely participate in the full phenotyping protocol. All others will be contacted by the protocol team to review exclusion criteria. Eligible patients will be invited to Clinical Research Center for a screening visit.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: men and women 18 years old and over with BMI > 30 BMI > 25 and < 30 BMI > 18.5 and < 25
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2007-03-08 (Actual)

PRIMARY OUTCOMES:
Phenotype (physical and behavioral traits) of overweight and obese people | Two weeks
  The aim of this study is to extensively phenotype subjects with varying degrees of obesity, as well as those with rare adipose disorders such as multiple symmetric lipomatosis (Madelung s disease), Dercums disease (adiposis dolorosa) and lipedema; to assess their hormonal, metabolic, cognitive and behavioral traits.

CONTACTS AND LOCATIONS:
Overall Officials: Ranganath Muniyappa, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adams KF, Schatzkin A, Harris TB, Kipnis V, Mouw T, Ballard-Barbash R, Hollenbeck A, Leitzmann MF. Overweight, obesity, and mortality in a large prospective cohort of persons 50 to 71 years old. N Engl J Med. 2006 Aug 24;355(8):763-78. doi: 10.1056/NEJMoa055643. Epub 2006 Aug 22. PMID 16926275
- [Background] Calle EE, Rodriguez C, Walker-Thurmond K, Thun MJ. Overweight, obesity, and mortality from cancer in a prospectively studied cohort of U.S. adults. N Engl J Med. 2003 Apr 24;348(17):1625-38. doi: 10.1056/NEJMoa021423. PMID 12711737
- [Background] Fontaine KR, Redden DT, Wang C, Westfall AO, Allison DB. Years of life lost due to obesity. JAMA. 2003 Jan 8;289(2):187-93. doi: 10.1001/jama.289.2.187. PMID 12517229
- [Derived] Meral R, Malandrino N, Walter M, Neidert AH, Muniyappa R, Oral EA, Brown RJ. Endogenous Leptin Concentrations Poorly Predict Metreleptin Response in Patients With Partial Lipodystrophy. J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1739-e1751. doi: 10.1210/clinem/dgab760. PMID 34677608
- [Derived] Armiyaw L, Sarcone C, Fosam A, Muniyappa R. Increased beta-Cell Responsivity Independent of Insulin Sensitivity in Healthy African American Adults. J Clin Endocrinol Metab. 2020 Jul 1;105(7):e2429-38. doi: 10.1210/clinem/dgaa234. PMID 32382759
- [Derived] Fosam A, Sikder S, Abel BS, Tella SH, Walter MF, Mari A, Muniyappa R. Reduced Insulin Clearance and Insulin-Degrading Enzyme Activity Contribute to Hyperinsulinemia in African Americans. J Clin Endocrinol Metab. 2020 Apr 1;105(4):e1835-46. doi: 10.1210/clinem/dgaa070. PMID 32052016
- [Derived] Kassai A, Muniyappa R, Levenson AE, Walter MF, Abel BS, Ring M, Taylor SI, Biddinger SB, Skarulis MC, Gorden P, Brown RJ. Effect of Leptin Administration on Circulating Apolipoprotein CIII levels in Patients With Lipodystrophy. J Clin Endocrinol Metab. 2016 Apr;101(4):1790-7. doi: 10.1210/jc.2015-3891. Epub 2016 Feb 22. PMID 26900642
- [Derived] Muniyappa R, Noureldin R, Ouwerkerk R, Liu EY, Madan R, Abel BS, Mullins K, Walter MF, Skarulis MC, Gharib AM. Myocardial Fat Accumulation Is Independent of Measures of Insulin Sensitivity. J Clin Endocrinol Metab. 2015 Aug;100(8):3060-8. doi: 10.1210/jc.2015-1139. Epub 2015 May 28. PMID 26020762
- [Derived] Muniyappa R, Sable S, Ouwerkerk R, Mari A, Gharib AM, Walter M, Courville A, Hall G, Chen KY, Volkow ND, Kunos G, Huestis MA, Skarulis MC. Metabolic effects of chronic cannabis smoking. Diabetes Care. 2013 Aug;36(8):2415-22. doi: 10.2337/dc12-2303. Epub 2013 Mar 25. PMID 23530011
- [Derived] Heikens MJ, Gorbach AM, Eden HS, Savastano DM, Chen KY, Skarulis MC, Yanovski JA. Core body temperature in obesity. Am J Clin Nutr. 2011 May;93(5):963-7. doi: 10.3945/ajcn.110.006270. Epub 2011 Mar 2. PMID 21367952
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2007-DK-0077.html